CLINICAL TRIAL: NCT02344446
Title: Physical Therapy Intervention for Extended Physical Symptoms After a Sports-related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walsh University (Other)
Responsible Party: Principal Investigator, Jennifer Reneker, Assistant Professor, Walsh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WalshU
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Concussion; Dizziness
Keywords: physical therapy intervention
MeSH Terms: conditions — Brain Concussion; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skilled Therapy (Experimental): Differential physical therapy treatment, based on assessment results, with follow-up visits for PT treatment 1 - 2 times per week until patient achieves at least 1 primary outcome. They will pragmatically design an individualized and progressive treatment plan, including manual therapy (manipulation and/or mobilization), neuromotor control strategies, and vestibular rehabilitation techniques, depending on the findings at assessment and patient response. Therapists can also tailor education regarding mental and physical rest according to specific parameters provided by the treating physician. Patients may also be prescribed a home exercise program and exercise education. The precise treatment strategies will be recorded.
  Interventions: Other: Skilled Therapy

INTERVENTIONS:
Other: Skilled Therapy — Active physical therapy treatment

SUMMARY:
The purpose of this study is to investigate if skilled physical therapy treatment for dizziness after sports-related concussion, delivered after greater than 30 days post-concussion is effective to remediate physical symptoms. This will be the first study that explores differential PT treatment for dizziness in concussed athletes who have physical symptoms 30+ days after concussion. The findings of this important research have great potential to influence clinical practice and place increased emphasis on and acceptance of manual skills and neuromotor training in the treatment of concussed patients with dizziness.

DETAILED DESCRIPTION:
Patients will be recruited from the ongoing Randomized Clinical Trial (Walsh University HSR 14-20) that are not returned to play and/or are not asymptomatic at the completion of their involvement in this research protocol. Based on the timeframe for their participation in the aforementioned study, these athletes will be 30 - 50 days post-concussion. At their final visit for the RCT, patients with one of the following criteria will be invited to participate in this research study:

1. Lack of release for Return to Play
2. Continuation of physical symptoms (headache, nausea, vomiting, balance problems, dizziness, light or noise sensitivity, numbness and/or vision problems) as recorded on the Post-Concussion Symptom Scale.

Desired sample size: 15 participants.

Skilled treatment: patients will be scheduled for a physical therapy assessment. The PTs will use a prescriptive approach to the assessment of the central nervous system, the cervical spine, and the vestibular system to determine the relative involvement of each system and dysfunction contributing to the patient's physical complaints. This assessment will include the outcome measures that will be obtained pre and post-treatment (Vertigo Symptom Scale (VSS) and the Functional Gait Assessment (FGA). Once the assessment is completed, the PT will initiate treatment, with follow-up visits for PT treatment 1 - 2 times per week. They will pragmatically design an individualized and progressive treatment plan, including manual therapy (manipulation and/or mobilization), neuromotor control strategies, and vestibular rehabilitation techniques, depending on the findings at assessment and patient response. Therapists can also tailor education regarding mental and physical rest according to specific parameters provided by the treating physician. Patients may also be prescribed a home exercise program and exercise education. The precise treatment strategies will be recorded. At each PT visit, symptomatic recovery will be tracked using the PCS.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the ongoing Randomized Clinical Trial (Walsh University HSR 14-20) that are not returned to play and/or are not asymptomatic at the completion of their involvement in this research protocol. Based on the timeframe for their participation in the aforementioned study, these athletes will be 30 - 50 days post-concussion. At their final visit for the RCT, patients with one of the following criteria will be invited to participate in this research study:

  1. Lack of release for Return to Play
  2. Continuation of physical symptoms (headache, nausea, vomiting, balance problems, dizziness, light or noise sensitivity, numbness and/or vision problems) as recorded on the Post-Concussion Symptom Scale

Exclusion Criteria:

* Any one who is not enrolled in the aforementioned RCT

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic Recovery | Within 6 months of enrollment
  Using the Post-Concussion Symptom Scale, self-reported symptomatic presentation will be tracked at each visit
Return to Play | Within 6 months of enrollment
  The treating physician will determine when return to play should be initiated.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Reneker, MSPT, Principal Investigator — Walsh Unviersity
Locations (1):
- Walsh University, North Canton, Ohio, United States